CLINICAL TRIAL: NCT04037800
Title: Impact of Sustainable Functional Urethral Reconstruction on Early Continence Recovery After Robotic-assisted Radical Prostatectomy: a Randomized Controlled Trial
Brief Title: An RCT to Compare Early Continence Recovery After RARP With or Without Sustainable Functional Urethral Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Yinghao Sun, Chief Physician, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CH-URO2019001
Record Dates: First submitted 2019-07-24; First posted 2019-07-30 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer; Urinary Incontinence
Keywords: Prostate cancer; Prostatectomy; Robotic surgery; Urinary incontinence; Sustainable functional urethral reconstruction
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SFUR-RARP (Experimental): Patients in which RARP with sustainable functional urethral reconstruction (SFUR) is performed.
  Interventions: Procedure: SFUR-RARP
- Standard RARP (Active Comparator): Patients in which standard RARP is performed.
  Interventions: Procedure: Standard RARP

INTERVENTIONS:
Procedure: SFUR-RARP — Robotic-assisted radical prostatectomy with sustainable functional urethral reconstruction (SFUR)
  Arms: SFUR-RARP
Procedure: Standard RARP — Robotic-assisted radical prostatectomy with conventional RARP procedures.
  Arms: Standard RARP

SUMMARY:
The study is a prospective randomized controlled trail to compare early urinary continence recovery after robotic-assisted radical prostatectomy with or without sustainable functional urethral reconstruction (SFUR).

DETAILED DESCRIPTION:
Early urinary incontinence has always been a tricky problem for both patients and urologists, even though over 90% patients can recover 1 year after surgery. Many urologists are trying to modify the surgical technique to resolve this problem. Sustainable functional urethral reconstruction (SFUR) is a novel technique which may improve early urinary continence recovery for both local and locally advanced prostate cancer, and even for those with high volume prostate by providing adequate urethral length with bladder neck tubularization and making sustainable periurethral support with peritoneal flap. The purpose of this study is to verify the impact of this new technique on early recovery of urinary continence, as well as on urinary function and oncological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥40, but ≤75 years old；
* Histological confirmed prostate cancer；
* Localized or locally advanced prostate cancer；
* Presence of urinary continence prior to the procedure;
* Informed consent signed;

Exclusion Criteria:

* Metastatic prostate cancer confirmed by ECT, PSMA or whole-body MRI;
* Presence of any prostatic surgery(such as transurethral resection, laser therapy, microwave therapy, radiofrequency ablation and so on) prior to the procedure;
* Radiation therapy of the prostate or pelvis prior to the procedure;
* Uncontrolled intercurrent illness that would limit compliance with study requirements;
* Any condition that contraindicates a radical prostatectomy;

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-12-08 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
1-month urinary continence recovery rates | 1 month after catheter removal
  Continence defined as daily usage of 0-1 pad with 24-hour pad weights≤50g.

SECONDARY OUTCOMES:
Short-term urinary continence recovery | Within 3 month after catheter removal
  Two definitions of urinary continence: daily usage of 0-1 pad with 24-hour pad weights gain≤50g, 0 pads per day. Besides, quantification of urine leakage with 24-hour pad weight.
Peri and postoperative complications | 1-year follow up
  Clavien-Dindo classification.
Post-operative oncological outcomes | 1-year follow up
  Two assessment methods: positive surgical margin (PSM) rates and 1-year biochemical recurrence-free survival (BFS, defined as two consecutive PSA levels>0.2 ng/mL).
Short-term urinary function and urinary function-related quality of life | 1-week, 2-week, 1-month, 3-month after catheter removal.
  International Prostatic Symptom Score(IPSS) and the IPSS quality of life score.

OTHER OUTCOMES:
1-year urinary continence recovery | 1-year from the intervention
  Two definitions of urinary continence: daily usage of 0-1 pad with 24-hour pad weights gain≤50g, 0 pads per day.
1-year urinary function and urinary function-related quality of life | 1-year from the intervention
  International Prostatic Symptom Score(IPSS) and the IPSS quality of life score.
Evaluation of urinary continence with ICIQ-UI-SF | 1-week, 2-week, 1-month, 3-month after catheter removal
  International Consultation on Incontinence Questionnaire-Urinary Incontinence-Short Form (ICIQ-UI-SF).
Post-operative sexual function | 1-year from the intervention
  Sexual Health Inventory for Men (SHIM) score >=17.

CONTACTS AND LOCATIONS:
Overall Officials: Yinghao Sun, MD, PHD, Study Chair — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ficarra V, Novara G, Rosen RC, Artibani W, Carroll PR, Costello A, Menon M, Montorsi F, Patel VR, Stolzenburg JU, Van der Poel H, Wilson TG, Zattoni F, Mottrie A. Systematic review and meta-analysis of studies reporting urinary continence recovery after robot-assisted radical prostatectomy. Eur Urol. 2012 Sep;62(3):405-17. doi: 10.1016/j.eururo.2012.05.045. Epub 2012 Jun 1. PMID 22749852
- [Background] Dev HS, Sooriakumaran P, Srivastava A, Tewari AK. Optimizing radical prostatectomy for the early recovery of urinary continence. Nat Rev Urol. 2012 Jan 24;9(4):189-95. doi: 10.1038/nrurol.2012.2. PMID 22270136
- [Background] Bessede T, Sooriakumaran P, Takenaka A, Tewari A. Neural supply of the male urethral sphincter: comprehensive anatomical review and implications for continence recovery after radical prostatectomy. World J Urol. 2017 Apr;35(4):549-565. doi: 10.1007/s00345-016-1901-8. Epub 2016 Aug 2. PMID 27484205
- [Background] Pavlovich CP, Rocco B, Druskin SC, Davis JW. Urinary continence recovery after radical prostatectomy - anatomical/reconstructive and nerve-sparing techniques to improve outcomes. BJU Int. 2017 Aug;120(2):185-196. doi: 10.1111/bju.13852. Epub 2017 Apr 17. PMID 28319318
- [Background] Bianchi L, Turri FM, Larcher A, De Groote R, De Bruyne P, De Coninck V, Goossens M, D'Hondt F, De Naeyer G, Schatteman P, Mottrie A. A Novel Approach for Apical Dissection During Robot-assisted Radical Prostatectomy: The "Collar" Technique. Eur Urol Focus. 2018 Sep;4(5):677-685. doi: 10.1016/j.euf.2018.01.004. Epub 2018 May 7. PMID 29402756